CLINICAL TRIAL: NCT03659513
Title: Pharmacokinetics of the Drugs and Their Biological Response in ECMO Patients
Brief Title: The Effect of ECMO on the Pharmacokinetics of the Drugs and Their Clinical Efficacy
Acronym: ECMOPK
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 825636
Record Dates: First submitted 2018-03-15; First posted 2018-09-06 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hypoxia; Extracorporeal Membrane Oxygenation Complication
Keywords: Hypoxia; ECMO; Antibiotics; Pharmacokinetics
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Enrolled subjects will have blood samples taken just before antibiotics transfusion, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 24 hours after routine administration of the drug in question. Each sample will be about 1-2 mL, for a total of about 12 mL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will examine the pharmacokinetics of the various, routinely given antibiotics, sedatives, and opioids in patients undergoing venous-venous extra-corporal oxygenation (ECMO). Little is known about the distribution and effectiveness of antibiotics in this particular patient population.

DETAILED DESCRIPTION:
Patients with severe hypoxia that is refractory to traditional therapies are occasionally placed on venous-venous extracorporal membrane oxygenation (vv ECMO) to provide a bridge during the time when lungs alone cannot provide necessary support. This procedure is gaining prominence but it is largely unknown how medications, especially antibiotics, given to the patient on ECMO is distributed throughout the body as compared to patients without ECMO. Since the serum level of medication determines the biological activity of the drug, it is important to know if there is a difference in drug distribution between ECMO and non-ECMO patients. The investigator already collected well-established data on several antibiotics on non-ECMO as a part of FDA labeling. The study will help to determine if the concentration of currently prescribed are sufficient enough to reach their intended concentration in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with respiratory failure undergoing ECMO.

Exclusion Criteria:

* Lack of consent
* Age less than 18 years old
* Hematocrit lower than 7

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing ECMO will be invited to participate. In order to determine pharmacokinetics of the drugs, the investgators need at least 10-15 subjects in order to create a pharmacological model. Since the site plan to study 3 antibiotics, propofol and hydromorphone, the investigators calculated the initial sample size at 50
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2016-09-13 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of the antibiotics - Maximal Serum Antibiotic Concentration | 24 hours
  The primary outcome is the data describing the Maximal Serum Antibiotic Concentration (Cmax) of the antibiotics after the onset of infusion.This will be achieved by serial measurements of the serum antibiotic levels at discrete time points for total of 24 hours after starting antibiotics. We will calculate Cmax to demonstrate maximal concentration of the antibiotics.
Pharmacokinetics of the antibiotics - Area Under Curve (AUC) | 24 hours
  The primary outcome is the data describing the Area Under Curve (AUC) of the antibiotics after the onset of infusion. This will be achieved by serial measurements of the serum antibiotic levels at discrete time points for total of 24 hours after starting antibiotics. We will calculate AUC to further demonstrate the distribution of antibiotic patients undergoing ECMO treatment.

SECONDARY OUTCOMES:
Clinical effectiveness of antibiotic dosing for ECMO patients | 3 months
  The investigators will correlate serum concentration of antibiotics to the resolution of infection, pressor requirements, and survival in patients. The surveillance will take place up to 3 months after the conclusion of the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Gutsche, MD, Principal Investigator — University of Pennsylvania; Krzysztof Laudanski, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States